CLINICAL TRIAL: NCT02469818
Title: Diagnostic Accuracy of Bedside Point of Care Ulrasound (POCUS) in the Management of the Shoulder Dislocations
Brief Title: Diagnostic Accuracy of Bedside Ultrasonography in the Management of the Shoulder Dislocations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaTRH005
Record Dates: First submitted 2015-06-08; First posted 2015-06-12 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Shoulder Dislocation
Keywords: pocus; ultrasonography; glenohumeral dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Shoulder dislocation is a common clinical presentation in the emergency department, comprising about 50 percent of all major joint dislocations. In the standart management of shoulder dislocations physicians generally need to see pre and post reduction x ray graphics. Ultrasonography is harmless way of evaluating shoulder and may be used in the management of the shoulder dislocations instead of the x ray evaluations.

DETAILED DESCRIPTION:
Shoulder dislocation is a common clinical presentation in the emergency department, comprising about 50 percent of all major joint dislocations. In the standard management of shoulder dislocations physicians generally need to see pre and post reduction x ray graphics. Ultrasonography is harmless way of evaluating shoulder and may be used in the management of the shoulder dislocations instead of the x ray evaluations.Recent literature has demonstrated the superiority of point-of-care ultrasonography (POCUS) in detecting both anterior and posterior shoulder dislocations, making it another rapidly evolving tool to improve accuracy, decrease error, and improve efficiency. The aim of the study is to evaluate the accuracy and clinical usability of ultrasonography in the management of the shoulder dislocations.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 14 years with suspected shoulder dislocation
* Accept to be participating

Exclusion Criteria:

* Patients under 15 years of age
* Diagnosed before pocus evaluation
* Open fracture dislocations of the shoulder

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients over 14 years of age with the complaint of shoulder pain and suspected glenohumeral dislocations
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of emergency physician performed point of care ultrasonography of shoulder in diagnosing of shoulder dislocations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Can K. Akyol, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Can K. Akyol, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Abbasi S, Molaie H, Hafezimoghadam P, Zare MA, Abbasi M, Rezai M, Farsi D. Diagnostic accuracy of ultrasonographic examination in the management of shoulder dislocation in the emergency department. Ann Emerg Med. 2013 Aug;62(2):170-5. doi: 10.1016/j.annemergmed.2013.01.022. Epub 2013 Mar 13. PMID 23489654
- [Background] Mackenzie DC, Liebmann O. Point-of-care ultrasound facilitates diagnosing a posterior shoulder dislocation. J Emerg Med. 2013 May;44(5):976-8. doi: 10.1016/j.jemermed.2012.11.080. Epub 2013 Mar 13. PMID 23490112
- [Background] Kahn JH, Mehta SD. The role of post-reduction radiographs after shoulder dislocation. J Emerg Med. 2007 Aug;33(2):169-73. doi: 10.1016/j.jemermed.2007.01.003. Epub 2007 Jun 13. PMID 17692769
- [Background] Hendey GW. Necessity of radiographs in the emergency department management of shoulder dislocations. Ann Emerg Med. 2000 Aug;36(2):108-113. doi: 10.1067/mem.2000.108314. PMID 10918101
- [Background] Gupta H, Robinson P. Normal shoulder ultrasound: anatomy and technique. Semin Musculoskelet Radiol. 2015 Jul;19(3):203-11. doi: 10.1055/s-0035-1549315. Epub 2015 May 28. PMID 26021582
- [Background] Smith MJ, Rogers A, Amso N, Kennedy J, Hall A, Mullaney P. A training, assessment and feedback package for the trainee shoulder sonographer. Ultrasound. 2015 Feb;23(1):29-41. doi: 10.1177/1742271X14566067. PMID 25866545
- [Derived] Akyol C, Gungor F, Akyol AJ, Kesapli M, Guven R, Cengiz U, Toksul HI, Eken C. Point-of-care ultrasonography for the management of shoulder dislocation in ED. Am J Emerg Med. 2016 May;34(5):866-70. doi: 10.1016/j.ajem.2016.02.006. Epub 2016 Feb 16. PMID 26935225